CLINICAL TRIAL: NCT04634045
Title: Targeting Self-Regulation in Family-Based Behavioral Treatment for Obesity and Cardiovascular Disease Prevention
Brief Title: Virtual Health Focused Acceptance-Based Program for Parents and Youth
Acronym: vHAPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Childrens of Alabama Kaul Pediatric Research Institute (Unknown)
Responsible Party: Principal Investigator, Marissa Gowey, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300005967
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Obesity; Executive Function
Keywords: Pediatric Obesity; Executive Function; Behavioral Intervention; Acceptance Based
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-Based Treatment (Experimental): A web-based treatment for pediatric overweight or obesity will be piloted with 10 caregiver and child pairs. Assessments will take place pre (0 months), post intervention (3.5 months) and at six months post-intervention (9.5 months) to evaluate patient outcomes, acceptability and feasibility.
  Interventions: Behavioral: Web Based Treatment

INTERVENTIONS:
Behavioral: Web Based Treatment — The literature regarding the efficacy of web-based platforms for behavioral weight management interventions in pediatric populations continues to grow. Considering the continued increase in technology and internet use among youth, web-based interventions have the potential to serve as a more cost-effective and personalized approach to pediatric behavioral weight management. Extant research supports this consideration. More research that compares web-based vs. traditional delivery of acceptance-based pediatric behavioral weight management interventions is necessary to understand the utility of this platform as well as which aspects are most effective.
  Other Names: Acceptance-Based Treatment

SUMMARY:
The main purpose of vHAPPY is to pilot test a new type of virtual family-based healthy lifestyle program for children aged 8-14 with obesity and their caregivers. vHAPPY aims to (1) Transition a previously developed acceptance-based behavioral treatment to web-based platform, utilizing qualitative and quantitative program evaluation data from past participants. (2) Determine the feasibility, acceptability, and preliminary outcomes of the adapted web-based treatment. (3) Evaluate whether the adapted web-based treatment (self-guided treatment + brief coaching) is similar to the traditional treatment (interventionist-guided treatment) in terms of feasibility, acceptability, and preliminary outcomes utilizing a non-randomized sequential arm design.

DETAILED DESCRIPTION:
Caregiver and child pairs will complete a 14 week virtual, self-guided healthy lifestyle program including education on health and wellness topics such as food groups, physical activity and stress management. Special skill builders for managing the thoughts, feelings and emotions associated with changing health behaviors will also be included. Pairs will have biweekly 15 minute coaching sessions to check in on progress in the past week, set goals and problem solve. Optional group sessions will be offered for peer support. In order to assess progress, pairs will also complete assessment visits before and after the program. These visits include one virtual assessment via Zoom and one in-person assessment at the University of Alabama at Birmingham. Caregivers and children will complete questionnaires and measures such has height, weight, blood pressure and a finger prick.

ELIGIBILITY:
Inclusion Criteria:

Children who:

1. have a BMI ≥ 85th percentile;
2. are 8 and 14 years old at the beginning of treatment;
3. can read, write, and speak English, along with their caregiver;
4. plan to stay living in the local area during the study period;
5. have a consenting caregiver who can commit to all study procedures.

Exclusion Criteria:

Children who:

1. have been diagnosed with a medical condition and/or are taking medication known to affect appetite/weight, physical activity level or executive function;
2. are currently participating in a formal weight management program beyond usual medical care or have a caregiver participating in a formal weight management program.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability - Interviews | 3.5 months
  Semi-structured group interviews will assess caregiver and child experiences with the program.
Acceptability - Surveys | 3.5 months
  Surveys will assess the utility of intervention content, intervention burden and satisfaction, participation barriers, and suggestions for change.
Feasibility - Interviews | 3.5 months
  Semi-structured group interviews will assess caregiver and child experiences with the program.
Feasibility - Surveys | 3.5 months
  Surveys will assess the utility of intervention content, intervention burden and satisfaction, participation barriers, and suggestions for change.

SECONDARY OUTCOMES:
Child Body Mass Index Z-Score | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Measure child's height and weight. Enter into the Children's Hospital Of Philadelphia Body Mass Index calculator.
Parent Body Mass Index | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Measure parent's height and weight. Enter into the Centers for Disease Control adult Body Mass Index calculator.
Parent Subjective Executive Function | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Behavior Rating Inventory of Executive Function (BRIEF) - Adult. Subjective EF will be measured using the Behavioral Rating Inventory of Executive Function. The Global Severity Index will be used which is interpreted using T-scores. Higher t-scores indicate better function.
Child Subjective Executive Function | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Behavior Rating Inventory of Executive Function (BRIEF) screener and BRIEF 2 (parent-report). Subjective EF will be measured using the Behavioral Rating Inventory of Executive Function. The Global Severity Index will be used which is interpreted using T-scores. Higher t-scores indicate better function.
Parent Behavioral Functioning - Anxiety | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Generalized Anxiety Disorder 7. Self-report questionnaire that will be used to measure parent anxiety symptoms over the past 2 weeks. Responses are coded 0-3. 0 = Not at all and 3 = Nearly every day. Total scores range from 0-21 and are ranked from minimal anxiety to severe anxiety.
Parent Behavioral Functioning - Depression | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Patient Health Questionnaire 8. Self-report questionnaire that will be used to measure parent depressive symptoms over the past 2 weeks. Eight items, each of which is scored 0-3, providing a 0-24 severity score.
Child Behavioral Functioning - Overall | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Pediatric Symptom Checklist -17. A parent-proxy report screener of child risk for internalizing (depression), externalizing (oppositional defiant disorder), and attention problems (ADHD). Each item is rated as never, sometimes or often present and scored 0,1 and 2 respectively. Total score is calculated by adding together the score for each item. Three subscale scores (attention, externalizing and internalizing) are calculated by adding the score for appropriately categorized items.

OTHER OUTCOMES:
Child Physical Activity Behavior | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Physical Activity Questionnaire - Child. A self-administered, 7 day recall instrument developed to assess general levels of physical activity in children approximately 8-14 years of age. Provides a summary physical activity score derived from nine items, each scored on a 5 point scale.
Child Eating Behavior | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Children's Eating Behavior Questionnaire. A 35-item parent proxy-report measure of eating behavior producing 8 subscales: responsiveness to food, enjoyment of food, satiety responsiveness, slowness in eating, fussiness, emotional overeating, emotional undereating, desire for drinks. Items are scored on a 5-point Likert scale and the mean score of each subscale is used. Higher scores indicate more eating behaviors in a certain domain.
Impact of the Food Environment | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Power of Food Scale. A 15-item self-report assessment of the psychological impact of living in food-abundant environments. Items are rated on a 5-point Likert scale and summed to create a total score. Higher scores reflect greater responsiveness to the food environment.
Child Psychological Flexibility - Acceptance | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Acceptance Fusion Questionnaire for Youth. A 17-item self-report measure for to assess psychological inflexibility in children. Items are scored on a 5-point Likert scale and summed for a total score ranging between 0-68. Higher scores are indicative of greater psychological inflexibility.
Child Psychological Flexibility - Mindfulness | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Child and Adolescent Mindfulness Measure. A 10-item measure of children's awareness and acceptance of their own private events or internal experiences. Items are reverse scored on a 5-point Likert scale. Higher scores correspond to higher levels of mindfulness.
Parent Psychological Flexibility | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Parental Acceptance and Action Questionnaire. A 15-item measure that evaluates parents' experiential acceptance and action tendencies in the context of their relationship with their children. The Total score is used which is a sum of all items which are rated on a 7-point Likert scale. Higher scores represent a greater degree of parental experiential avoidance.
Demographics | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Child and caregiver characteristics such as age, sex, race/ethnicity, educational level, family income, and marital status will be assessed via caregiver report.
Participant Satisfaction - Interviews | 3.5 months
  Semi-structured group interviews will assess caregiver and child experiences with the program.
Participant Satisfaction - Surveys | 3.5 months
  Surveys will assess the utility of intervention content, intervention burden and satisfaction, participation barriers, and suggestions for change.
Adherence | 3.5 months
  Number of Sessions Attended
Child Health Related Quality of Life - Self Report | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Sizing Me Up©. A validated obesity-specific self-report measure, respectively, of health-related quality of life for children 5-13 years old that measure functioning in a variety of areas (e.g., emotional, physical, teasing/marginalization). The Total Score will be used as the outcome, which is a scaled score ranging from 0-100 with higher scores representing better quality of life.
Child Health Related Quality of Life - Parent Report | Baseline (0 weeks), post intervention (14 weeks) and six months post intervention (38 weeks)
  Sizing Them Up©. A validated obesity-specific parent-report measure, respectively, of health-related quality of life for children 5-13 years old that measure functioning in a variety of areas (e.g., emotional, physical, teasing/marginalization). The Total Score will be used as the outcome, which is a scaled score ranging from 0-100 with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa A Gowey, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size and risk of confidentiality loss, there is no plan to share IPD.